CLINICAL TRIAL: NCT05642065
Title: Does a Hip Muscle Activation Home Exercise Program Change Patient Performance on the Forward Step-Down Test? A Single-Arm Clinical Trail
Brief Title: Hip Activation and FSDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Daniel W. Flowers, Assistant Professor of Physical Therapy, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002264
Record Dates: First submitted 2022-11-28; First posted 2022-12-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Movement, Abnormal; Lower Extremity Problem
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants will undergo lower extremity movement assessment on the Forward Step Down Test before and after a home exercise program (HEP) consisting of five hip activation exercises. These exercises will be performed 2x/week for 8 weeks. Surface EMG of the gluteus maximus and medius, in addition to tracking of participant compliance on the HEP program will also be assessed pre- and post-intervention.
  Interventions: Other: Hip muscle activation home exercise program

INTERVENTIONS:
Other: Hip muscle activation home exercise program — Participants will perform a home exercise program consisting of five hip muscle activation exercises with the use of a resistance band. The program will be eight weeks in duration, and participants will perform the exercises twice weekly.

SUMMARY:
The purpose of this study is to determine if activation training of the hip musculature affects muscle activation and frontal plane mechanics in healthy individuals.

Specific Aim 1: Determine whether performance on the forward step-down test (FSDT) changes after an eight-week home exercise program (HEP) focused on hip musculature activation in healthy individuals.

Specific Aim 2: Determine whether surface electromyography (sEMG) hip musculature changes following an eight-week HEP focused on hip musculature activation in healthy individuals.

Specific Aim 3: Determine whether a dose-response relationship exists between compliance on the HEP and changes in FSDT scores in healthy individuals.

Specific Aim 4: Determine whether a dose-response relationship exists between compliance on the HEP and sEMG changes in hip musculature activation in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be current first or second year Doctor of Physical Therapy students in the School of Allied Health Professions at LSU Health Shreveport.

Exclusion Criteria:

* Current knee pain or pathology in the dominant leg, and women with known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Scores on the Forward Step Down Test | Pre- and Post- Intervention Program (8 weeks)
  Participants will perform the Forward Step Down Test pre- and post-intervention, while being score by two investigators simultaneously.

SECONDARY OUTCOMES:
Surface electromyography (sEMG) - Gluteus Maximus | Pre- and Post- Intervention Program (8 weeks)
  sEMG data for the gluteus maximus, including both mean EMG activation and peak EMG activation will be recorded during performance of the Forward Step Down Test.
Surface electromyography (sEMG) - Gluteus Medius | Pre- and Post- Intervention Program (8 weeks)
  sEMG data for the gluteus medius, including both mean EMG activation and peak EMG activation will be recorded during performance of the Forward Step Down Test.
Home Exercise Program (HEP) Compliance | Pre- and Post- Intervention Program (8 weeks)
  Participants will complete a log of the number of HEP sessions they complete during the 8-week intervention program. The sum of sessions completed will be used as a measure of compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W. Flowers, DPT, PhD, Principal Investigator — Louisiana State University Health Sciences Center Shreveport
Locations (1):
- Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT05642065/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT05642065/ICF_001.pdf